CLINICAL TRIAL: NCT01756066
Title: A Test of Different Degrees of Cost Sharing on Program Uptake and Attendance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Harvard University (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 816444
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
Keywords: Obesity; Weight loss program; incentives
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Active Comparator): Participant has 50% subsidy, i.e. gets a 50% discount off regular price of the program
  Interventions: Behavioral: Different levels of cost sharing
- B (Experimental): Participant has 100% subsidy, i.e. program attendance is free
  Interventions: Behavioral: Different levels of cost sharing
- C (Experimental): Participant has 80% subsidy; i.e. gets 80% discount off regular price of the program
  Interventions: Behavioral: Different levels of cost sharing
- D (Experimental): Participant has 50% subsidy up front (i.e. pays 50%), with possibility for 100% subsidy based on attaining monthly participation goals
  Interventions: Behavioral: Different levels of cost sharing

INTERVENTIONS:
Behavioral: Different levels of cost sharing

SUMMARY:
To test the uptake of four different cost sharing discounts for enrolling in the Weight Watchers weight loss program as well as outcomes (program attendance and weight loss) over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Must be employee of Vanguard Health Systems over the age of 18
2. Must have a BMI of 21 or greater

Exclusion Criteria:

1. Must not be under the age of 18
2. Must not have a BMI lower than 21

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1239 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Uptake | 12 months
  the percent of patients who sign up for the program, by arm

SECONDARY OUTCOMES:
Efficacy | 12 months
  Program attendance and weight loss among participants who sign up for the program

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Ingersoll Rand, Davidson, North Carolina
  - Vanguard Health Systems, Nashville, Tennessee

REFERENCES:
- [Derived] John LK, Troxel AB, Yancy WS Jr, Friedman J, Zhu J, Yang L, Galvin R, Miller-Kovach K, Halpern SD, Loewenstein G, Volpp K. The Effect of Cost Sharing on an Employee Weight Loss Program: A Randomized Trial. Am J Health Promot. 2018 Jan;32(1):170-176. doi: 10.1177/0890117116671282. Epub 2016 Oct 21. PMID 29277125